CLINICAL TRIAL: NCT02800148
Title: Bioequivalence Study of Two Treatments in the Treatment of Inflammatory Lesions of Rosacea on the Face
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Collaborators: DPT Laboratories, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-16-009
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azelaic acid foam (Experimental)
  Interventions: Drug: Azelaic acid foam
- Finacea Foam (Active Comparator)
  Interventions: Drug: Azelaic acid foam
- Placebo Foam (Placebo Comparator)
  Interventions: Drug: Azelaic acid foam - Placebo

INTERVENTIONS:
Drug: Azelaic acid foam
  Arms: Azelaic acid foam
Drug: Azelaic acid foam
  Other Names: Finacea Foam
  Arms: Finacea Foam
Drug: Azelaic acid foam - Placebo
  Arms: Placebo Foam

SUMMARY:
To compare the bioequivalence of Perrigo's azelaic acid foam product to Finacea Foam for the treatment of Inflammatory Lesions of Rosacea

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign an Institutional Review Board (IRB) approved written informed consent for this study.
2. Subjects must be at least 18 years of age.
3. Subjects must have a definite clinical diagnosis of moderate to facial papulopustular rosacea,
4. Subjects must be willing and able to understand and comply with the requirements of the study, apply the medication as instructed, refrain from use of all other
5. Subjects must be in general good health and free from any clinically significant disease, other than rosacea, that might interfere with the study evaluations.
6. Females of childbearing potential (excluding women who are surgically sterilized (verified tubal ligation or bilateral oophorectomy or hysterectomy) or post- menopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day 1 (Baseline), must be willing to use an acceptable form of birth control during the study.

Exclusion Criteria:

1. Subjects, who are pregnant, breastfeeding, or planning a pregnancy within the period of their study participation.
2. Current or past ocular rosacea
3. Presence of any other facial skin condition that might interfere with rosacea diagnosis and/or assessment
4. Any uncontrolled, chronic or serious disease or medical condition that would prevent participation in a clinical trial or, in judgment of the Investigator, would put the subject at undue risk or might confound the study assessments
5. Currently using any product containing Azelaic Acid/or belonging to the same family as Azelaic Acid foam, 15%.
6. Any use of Azelaic Acid Foam, 15%, 1 month (30 days) prior to baseline or throughout the study.
7. History of hypersensitivity or allergy to Finacea® (Azelaic Acid) Foam, 15%, and/or any ingredient in the study medication.
8. Use of radiation therapy and/or anti-neoplastic agents within 90 days prior to Visit 1/Day 1 (Baseline).
9. Current use of anticoagulation therapy and use throughout the study.
10. Use of medicated make-up (including anti-aging make-up) throughout the study
11. Use during the study of 1) systemic steroids, 2) topical retinoids to the face 3) antibiotics known to impact rosacea 4) immunosuppressive agents, or immunomodulators).
12. Facial use of 1) topical steroids, 2) topical anti-inflammatory agents, 3) topical antimycotics, 4) any topical rosacea treatments or 4) topical antibiotics.
13. Use of medicated cleansers on the face throughout the study.
14. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements
15. Use of topical astringents or abrasives, medicated topical preparations (prescription and OTC products) within 2 days prior to Visit 1 and throughout the study.
16. Use of antipruritics (including antihistamines), spa treatments or chlorine exposure (swimming etc.) within 24 hours of all study visits.
17. Participation in any clinical study involving an investigational product, agent or device that might influence the intended effects or mask the side effects of study medication in the 1 month (30 days) prior Visit 1/Day 1 (Baseline) or throughout the study.
18. Previous enrollment in this study or current enrollment in this study at another participating site.
19. Use of tanning booths, sun lamps (excessive UV radiation e.g., phototherapy, daily extended exposure or occupational exposure to the sun), sunbathing or excessive exposure to the sun 1 week prior to baseline and throughout the study.
20. Subjects who in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consultants, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azelaic Acid Foam; Finacea Foam: Azelaic acid foam
- Placebo Foam: Azelaic acid foam - Placebo
Period: Overall Study
Arm/Group | Azelaic Acid Foam | Finacea Foam | Placebo Foam
Started | 224 | 224 | 219
Completed | 199 | 204 | 194
Not Completed | 25 | 20 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Foam | Finacea Foam | Placebo Foam | Total
Number analyzed (Participants) | 224 | 224 | 219 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (13.85) | 51.5 (13.67) | 49.0 (12.42) | 50.7 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 167 | 166 | 497
  Male | 60 | 57 | 53 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 55 | 68 | 183
  Not Hispanic or Latino | 164 | 169 | 151 | 484
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 4
  Asian | 1 | 5 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 221 | 215 | 211 | 647
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change (Reduction) of Lesion Count From Day 1
Time Frame: Day 84
Measure: Mean (Standard Deviation); unit: percentage of lesion reduction
Arm/Group | Azelaic Acid Foam | Finacea Foam | Placebo Foam
Number analyzed (Participants) | 178 | 181 | 178
percentage of lesion reduction | 61.14 (33.623) | 57.27 (34.513) | 49.43 (44.437)
Statistical Analysis 1: Comparison: Azelaic Acid Foam vs Finacea Foam; Test type: Equivalence — provides 85% power of success; Fieller's method — No p-value as calculated for bioequivalence, just a T/R ratio and 90% confidence interval; equivalence ratio = 107, 90% CI 2-sided [96.1 to 115.5]

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Azelaic Acid Foam | Finacea Foam | Placebo Foam
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/224 | 0/219
Serious Adverse Events (participants affected / at risk) | 1/224 | 0/224 | 2/219
Other Adverse Events (participants affected / at risk) | 0/224 | 0/224 | 0/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azelaic Acid Foam (N=224) | Finacea Foam (N=224) | Placebo Foam (N=219)
Esophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aseptic Meningitis (Infections and infestations) | 0 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's cannot disclose trial results under any circumstances.

DOCUMENTS (2):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02800148/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02800148/SAP_001.pdf